CLINICAL TRIAL: NCT00171015
Title: An Open,Multicenter Study to Evaluate the Efficacy and Safety of a 4 Week Therapy With Valsartan/Hydrochlorothiazide 160/25 (Fixed Dose Combination of Valsartan 160 mg Plus HCTZ 25 mg) in Patients Not Adequately Responding to a 4 Week Monotherapy With Olmesartan Medoxomil 40 mg or Combination Therapy With Olmesartan Medoxomil 20 mg Plus HCTZ 12.5 mg
Brief Title: VALORY Study of Valsartan/Hydrochlorizide for Patients Who do Not Respond Adequately to Olmesartan Medoxomil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAH631BDE10
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: VALSARTAN; HYDROCHLOROTHIAZIDE; OLMESARTAN; HYPERTENSION
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: valsartan plus hydrochlorothiazide

SUMMARY:
To evaluate the efficacy of valsartan 160 mg/HCTZ 25 mg in patients not adequately responding to monotherapy with olmesartan medoxomil 40 mg or combination therapy with olmesartan medoxomil 20 mg plus HCTZ 12.5 mg by testing the hypothesis that valsartan 160 mg/HCTZ 25 mg significantly reduces the trough mean sitting diastolic blood pressure (MSDBP) after a 4-week treatment in the nonresponder population.

ELIGIBILITY:
Inclusion Criteria:

* Females must be either post-menopausal for one year, surgically sterile or using effective contraceptive methods (e.g. barrier method with spermicide, intra-uterine device, hormonal contraceptives).
* Patients with essential hypertension:

  * At Visit 1, untreated patients should have a MSDBP >100 mmHg and < 110 mmHg and treated patients need to have a MSDBP < 110 mmHg. Untreated patients can be included as soon as the safety laboratory parameters are available, but not at the day of Visit 1. This inclusion visit will be recorded as Visit 3 in the CRF.
  * At Visit 2, patients previously treated for hypertension need to have a MSDBP ≥ 100 mmHg and < 110 mmHg for entrance into the first treatment phase. Patients previously treated for hypertension who have a MSDBP < 100 mmHg at Visit 2 will continue the wash-out phase and will be again evaluated with regard to BP criteria at Visit 3. Untreated patients do not perform Visit 2.
  * At Visit 3, which is not performed for patients who entered the first treatment phase already at Visit 2, patients need to have a MSDBP >100 mmHg and < 110 mmHg for entrance into the first treatment phase.
  * At Visit 4, all patients need to have a MSDBP >90 mmHg for entrance into the second treatment phase.

Exclusion Criteria:

* MSDBP >110 mmHg or MSSBP >180 mmHg
* Pregnant or nursing women
* Inability to completely discontinue all antihypertensive medications safely for a period of up to 2 weeks, as required by the protocol

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2004-12; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 4 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 4 weeks
Diastolic blood pressure less than 90 mmHg after 4 weeks
Diastolic blood pressure less than 90 mmHg or decrease in diastolic blood pressure of 10 mmHg or greater after 4 weeks
Change from baseline heart rate after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Multiple Locations, Germany
- Novartis Pharmaceuticals, Basel, Switzerland